CLINICAL TRIAL: NCT01292863
Title: The Impact of a Biocompatible Peritoneal Dialysis Solution (Delflex Neutral pH) on Mesothelial Cell Viability and Peritoneal Transport
Brief Title: The Impact of Delflex on Mesothelial Cell Viability and Peritoneal Transport
Acronym: Delflex
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was modified to in vitro design and no longer involves participants
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Fresenius Medical Care North America (Industry)
Responsible Party: Principal Investigator, Cindy Denu-Ciocca, MD, Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-2359
Record Dates: First submitted 2011-02-08; First posted 2011-02-10 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-02

CONDITIONS: End Stage Renal Disease
Keywords: Peritoneal dialysis; Biocompatible dialysis fluid
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Conventional peritoneal dialysis solution (Active Comparator): Subjects will be randomized to perform dialysis with the conventional peritoneal dialysis solution for 3 months. At the end of three months mesothelial cell shedding and apoptosis will be measured.
  Interventions: Other: Active Comparator: Conventional peritoneal dialysis solution
- Novel biocompatible dialysis solution Delflex neutral pH (Experimental)
  Interventions: Other: Experimental: Novel biocompatible dialysis solution

INTERVENTIONS:
Other: Active Comparator: Conventional peritoneal dialysis solution — Daily dialysis solution to be used for 3 months in crossover fashion.
  Other Names: Delflex
  Arms: Conventional peritoneal dialysis solution
Other: Experimental: Novel biocompatible dialysis solution — Daily dialysis solution to be used for 3 months in crossover fashion.
  Other Names: Delflex neutral pH
  Arms: Novel biocompatible dialysis solution Delflex neutral pH

SUMMARY:
The purpose of this study is to evaluate the impact of Delflex neutral pH (a biocompatible peritoneal dialysis solution) on mesothelial cell viability and peritoneal transport.

DETAILED DESCRIPTION:
In spite of its benefits, many peritoneal dialysis patients ultimately have to switch dialysis therapy to hemodialysis secondary to technique failure. Numerous etiologies for peritoneal dialysis treatment failure exist and include the continuous exposure of the peritoneal membrane to bioincompatible dialysis solutions with acidic pH and high content of glucose degradation products. These factors have been implicated in mesothelial cell loss, fibrosis and neovascularization, resulting in alterations in solute transport and ultrafiltration failure. Novel peritoneal dialysis solutions with neutral pH and low concentrations of glucose degradation products have recently been developed to improve biocompatibility and ameliorate the consequences of membrane damage with conventional peritoneal dialysis solutions. While novel peritoneal dialysis solutions have been available outside the United States for several years, Delflex Neutral pH has only recently been approved for use in the United States. Thus, the majority of all the data supporting the benefits of these novel solutions comes from locations outside of the United States.

The central question regarding the novel peritoneal dialysis solution is whether long term use will result in better preservation of the peritoneal membrane to support dialysis. Ultimately, this can only be determined with studies comparing long term outcomes of patients using the various solutions. However, given the expected availability in the United States and the potential benefits of the novel peritoneal dialysis solutions long term studies comparing outcomes with conventional solutions raises ethical concerns. Therefore, surrogate markers for peritoneal membrane integrity are necessary. Short term studies using various surrogate markers to assess mesothelial cell mass and peritoneal inflammation such as Cancer Antigen 125 (CA125) and pro-inflammatory cytokines have been reported, but it is uncertain how well these markers predict long term outcome. Recently, a novel approach to predict outcome has been reported, using mesothelial cell shedding and apoptosis. The number of mesothelial cells and the number of apoptotic mesothelial cells in a standard 8 hour dialysis dwell were reported to correlate well with deterioration of peritoneal dialysis characteristics over a one year follow-up. The authors concluded that mesothelial cell shedding and apoptosis are reliable predictors of peritoneal membrane deterioration.

The purpose of this study is to evaluate the impact of Delflex neutral pH (a biocompatible peritoneal dialysis solution) on mesothelial cell viability and peritoneal transport. The study will specifically compare mesothelial cell shedding and apoptosis in the peritoneal dialysis effluent after exposure to Delflex neutral pH solution and conventional peritoneal dialysis solution. Cancer Antigen 125 (CA125)levels (indicative of mesothelial cell mass) and connective tissue growth factor (CTGF) levels (a marker of inflammation) will be measured in the spent dialysate to determine whether these markers correlate with cell shedding and apoptosis. The study will also characterize the transport of glucose degradation products (GDPs) and advanced glycosylation end products (AGEs) across the mesothelial cells after exposure to Delflex neutral pH solution versus conventional peritoneal dialysis solution.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age
* Incident or prevalent patients with End Stage Kidney disease treated with either CAPD (continuous ambulatory peritoneal dialysis) or CCPD (continuous cycling peritoneal dialysis)
* Patients must maintain modality of either CAPD or CCPD throughout duration of study
* Able to provide informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Recent (< 3 months) history of peritonitis
* CCPD utilizing Baxter cycler (due to inability to connect Delflex solution to cycler)
* Anticipated renal transplant within 6 months of enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-03; Primary Completion 2012-02 (Estimated); Study Completion 2012-05 (Estimated)

PRIMARY OUTCOMES:
Mesothelial cell shedding and apoptosis | 6 months
  Mesothelial cell shedding has been recently reported to predict deterioration of the peritoneal membrane.The novel peritoneal dialysis solution, Delflex neutral pH solution may decrease peritoneal inflammatory response resulting in less mesothelial cell shedding and apoptosis in the peritoneal dialysis effluent compared to use with standard peritoneal dialysate.
  The primary specific aim of the current project is to compare the effect of Delflex neutral pH solution with conventional dialysis solution on mesothelial cell shedding and apoptosis

SECONDARY OUTCOMES:
Cancer antigen 125 (CA 125) in spent dialysate | 6 months
  Cancer antigen 125 (CA 125) is a marker of mesothelial cell mass and studies have shown significantly increased levels of CA 125 utilizing novel biocompatible peritoneal dialysis solutions compared to conventional solutions. We plan to determine whether CA 125 correlate with effluent total and apoptotic mesothelial cells.
Characterize the mesothelial transport of glucose degradation products (GDPs) and advanced advanced glycosylation end products (AGEs) | 6 months
  Theoretically, a promising benefit of utilizing the novel peritoneal dialysis solutions is the beneficial effect of reduced local and systemic damage secondary to advanced glycosylation products. A recent study found a significant decrease in circulating AGE levels in patients treated with low GDP solution over 3 months compared to levels after 3 months using standard peritoneal dialysis fluid. We plan to characterize the mesothelial transport of GDPs and AGEs after exposure to Delflex neutral pH solution versus conventional peritoneal dialysis solution.
Connective tissue growth factor(CTGF)in spent dialysis fluid | 6 months
  Connective tissue growth factor (CTGF) levels in spent peritoneal dialysis fluid are strongly associated with high peritoneal solute transport rate and ultrafiltration failure. Connective tissue growth factor (CTFG) may be another marker of peritoneal membrane fibrosis and thus predictive of dialysis membrane failure. We plan to determine whether CTGF levels correlate with effluent total and apoptotic mesothelial cells.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia J Denu-Ciocca, MD, Principal Investigator — University of North Carolina, Chapel Hill

REFERENCES:
- [Background] Davies SJ, Russell L, Bryan J, Phillips L, Russell GI. Impact of peritoneal absorption of glucose on appetite, protein catabolism and survival in CAPD patients. Clin Nephrol. 1996 Mar;45(3):194-8. PMID 8706362
- [Background] Williams JD, Craig KJ, Topley N, Von Ruhland C, Fallon M, Newman GR, Mackenzie RK, Williams GT. Morphologic changes in the peritoneal membrane of patients with renal disease. J Am Soc Nephrol. 2002 Feb;13(2):470-479. doi: 10.1681/ASN.V132470. PMID 11805177
- [Background] Williams JD, Craig KJ, von Ruhland C, Topley N, Williams GT; Biopsy Registry Study Group. The natural course of peritoneal membrane biology during peritoneal dialysis. Kidney Int Suppl. 2003 Dec;(88):S43-9. doi: 10.1046/j.1523-1755.2003.08805.x. No abstract available. PMID 14870877
- [Background] Pajek J, Kveder R, Bren A, Gucek A, Ihan A, Osredkar J, Lindholm B. Short-term effects of a new bicarbonate/lactate-buffered and conventional peritoneal dialysis fluid on peritoneal and systemic inflammation in CAPD patients: a randomized controlled study. Perit Dial Int. 2008 Jan-Feb;28(1):44-52. PMID 18178947
- [Background] Williams JD, Topley N, Craig KJ, Mackenzie RK, Pischetsrieder M, Lage C, Passlick-Deetjen J; Euro Balance Trial Group. The Euro-Balance Trial: the effect of a new biocompatible peritoneal dialysis fluid (balance) on the peritoneal membrane. Kidney Int. 2004 Jul;66(1):408-18. doi: 10.1111/j.1523-1755.2004.00747.x. PMID 15200450
- [Background] Theodoridis M, Passadakis P, Kriki P, Gioka T, Panagoutsos S, Mourvati E, Thodis E, Kantartzi K, Vargemezis V. The alteration of dialysate cancer antigen 125 concentration under a biocompatible bicarbonate peritoneal dialysis solution and the preservation of the mesothelial cell viability. Ren Fail. 2008;30(2):161-7. doi: 10.1080/08860220701808384. PMID 18300115
- [Background] Kanjanabuch T, Siribamrungwong M, Khunprakant R, Kanjanabuch S, Jeungsmarn P, Achavanuntakul B, Pongpirul K, Park MS, Tungsanga K, Eiam-Ong S. Overnight mesothelial cell exfoliation: a magic tool for predicting future ultrafiltration failure in patients on continuous ambulatory peritoneal dialysis. Perit Dial Int. 2008 Jun;28 Suppl 3:S107-13. PMID 18552238
- [Background] Zarrinkalam KH, Stanley JM, Gray J, Oliver N, Faull RJ. Connective tissue growth factor and its regulation in the peritoneal cavity of peritoneal dialysis patients. Kidney Int. 2003 Jul;64(1):331-8. doi: 10.1046/j.1523-1755.2003.00069.x. PMID 12787426
- [Background] Mizutani M, Ito Y, Mizuno M, Nishimura H, Suzuki Y, Hattori R, Matsukawa Y, Imai M, Oliver N, Goldschmeding R, Aten J, Krediet RT, Yuzawa Y, Matsuo S. Connective tissue growth factor (CTGF/CCN2) is increased in peritoneal dialysis patients with high peritoneal solute transport rate. Am J Physiol Renal Physiol. 2010 Mar;298(3):F721-33. doi: 10.1152/ajprenal.00368.2009. Epub 2009 Dec 16. PMID 20015945
- [Background] Ishibashi Y, Sugimoto T, Ichikawa Y, Akatsuka A, Miyata T, Nangaku M, Tagawa H, Kurokawa K. Glucose dialysate induces mitochondrial DNA damage in peritoneal mesothelial cells. Perit Dial Int. 2002 Jan-Feb;22(1):11-21. PMID 11929138
- [Background] Morgan LW, Wieslander A, Davies M, Horiuchi T, Ohta Y, Beavis MJ, Craig KJ, Williams JD, Topley N. Glucose degradation products (GDP) retard remesothelialization independently of D-glucose concentration. Kidney Int. 2003 Nov;64(5):1854-66. doi: 10.1046/j.1523-1755.2003.00265.x. PMID 14531821
- [Background] Linden T, Forsback G, Deppisch R, Henle T, Wieslander A. 3-Deoxyglucosone, a promoter of advanced glycation end products in fluids for peritoneal dialysis. Perit Dial Int. 1998 May-Jun;18(3):290-3. PMID 9663893
- [Background] Thornalley PJ. Measurement of protein glycation, glycated peptides, and glycation free adducts. Perit Dial Int. 2005 Nov-Dec;25(6):522-33. PMID 16419322
- [Background] Li W, Hamada Y, Nakashima E, Naruse K, Kamiya H, Akiyama N, Hirooka H, Takahashi N, Horiuchi S, Hotta N, Oiso Y, Nakamura J. Suppression of 3-deoxyglucosone and heparin-binding epidermal growth factor-like growth factor mRNA expression by an aldose reductase inhibitor in rat vascular smooth muscle cells. Biochem Biophys Res Commun. 2004 Feb 6;314(2):370-6. doi: 10.1016/j.bbrc.2003.12.095. PMID 14733914